CLINICAL TRIAL: NCT05332834
Title: A Phase 1, First-in-Human, Double-Blind, Placebo-Controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SM17 When Administered Intravenously as a Single Ascending Dose in Healthy Subjects (Part A) and as Multiple Ascending Doses in Healthy Subjects (Part B)
Brief Title: A Phase 1 Study of Single and Multiple Intravenous Doses of SM17 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SinoMab BioScience Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM17-101
Record Dates: First submitted 2022-03-31; First posted 2022-04-18 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-02

CONDITIONS: Asthma
Keywords: SM17
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Biological Product: SM17 monoclonal antibody or Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug SM17 (Experimental): Peripheral intravenous injection
  Interventions: Biological: SM17
- Drug Placebo (Placebo Comparator): Peripheral intravenous injection
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: SM17 — Peripheral intravenous injection
  Arms: Drug SM17
Other: Placebo — Peripheral intravenous injection
  Arms: Drug Placebo

SUMMARY:
This trial is a phase 1, first-in-human, randomized, double-blind, placebo-controlled dose escalation trial following single and multiple doses intravenous administration of SM17.

It aims to evaluate the safety, tolerability, pharmacokinetic characteristics, pharmacodynamic effect and immunogenicity of single and multiple doses of SM17 injection in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfill all of the following inclusion criteria to be eligible for participation in the study:

1. Healthy, adult, male or female* (of non childbearing potential only), 19-55 years of age, inclusive, at the time of consent.

   * Females of non-childbearing potential are defined as follows:
   * Females who have undergone one of the following sterilization procedures at least 6 months prior to the first dosing:

     * Hysteroscopic sterilization.
     * Bilateral tubal ligation or bilateral salpingectomy.
     * Hysterectomy.
     * Bilateral oophorectomy or
   * Females who are postmenopausal with amenorrhea for at least 1 year prior to the first dosing and follicle stimulating hormone (FSH) serum levels consistent with postmenopausal status at the screening visit.
2. Male subjects must follow protocol specified contraception guidance as described in Section 12.4.5.
3. Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2 at the screening visit.
4. Is a non-smoker or ex-smoker who has stopped smoking for at least 6 months prior to the screening visit. Ex-smokers will have a history of <10 cigarettes pack-year.
5. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs (12-lead reporting RR, PR, QRS, QT and QTcF), as deemed by the PI or designee, at the screening visit and prior to the first dosing, including the following:

   * QTcF interval is ≤460 msec (males) and ≤470 msec (females) and has ECG findings considered normal or not clinically significant by the PI or designee.
6. Must sign an IRB-approved informed consent form (ICF) prior to any study-specific procedures.
7. Is able to comply with clinic visits and study-related procedures.

Exclusion Criteria:

Subjects must not be enrolled in the study if they meet any of the following criteria:

1. Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. History or evidence of a clinically significant disorder (including psychiatric), condition or disease that, in the opinion of the PI or designee would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.
3. History or current medical conditions, such as myocardial infarction or stroke within the 3 months prior to the screening visit, known cardiac disease, uncontrolled hypertension, and aortic or cerebral aneurysm.
4. Previously hospitalized for severe acute respiratory syndrome-coronavirus 2 (SARS Cov 2) prior to the screening visit.
5. Positive polymerase chain reaction test for SARS-CoV-2, either with the absence or presence of the clinical symptoms of COVID 19
6. Has evidence of any active or suspected bacterial, viral, fungal, or parasitic infections within the past 6 weeks prior to the screening visit (e.g., common cold, viral syndrome, flu-like symptoms). Subject who, in the opinion of the PI or designee, has a high risk of parasitic disease is also excluded.
7. Has known Type I/II diabetes.
8. Was vaccinated with live (attenuated) vaccinations within 1 month prior to the first dosing.
9. History of malignancy of any type, (with the exception of successfully treated in situ cervical cancer, or surgically excised non-melanomatous skin cancers) within 5 years prior to the screening visit.
10. History of any known primary or secondary immunodeficiency disorder.
11. History or presence of alcohol or drug abuse within the past 2 years prior to the first dosing.
12. Positive drugs and/or alcohol results at the screening visit or prior to the first dosing. Subject who has consumed alcohol within 48 hours prior to any study visit including the screening visit, will be excluded.
13. History or presence of hypersensitivity or idiosyncratic reaction to protein treatment, medications, any ingredients of SM17 or related compounds.
14. Female subjects of childbearing potential.
15. Female subject who is lactating or breastfeeding.
16. Female subject with a positive pregnancy test at the screening visit.
17. Has active infection including tuberculosis (TB) (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive hepatitis B surface antigen [HBsAg] result), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies). Subjects with a past or resolved hepatitis B virus infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Subjects positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA).
18. Uses of any over-the-counter or prescription medications (unless otherwise specified in this protocol) within the 14 days or 5 half-lives (whichever is longer), prior to receiving the first dose of SM17. Acetaminophen (up to 2 g per day) for analgesia, hormone replacement therapy (e.g., estrogen, thyroid), and spermicidal agents will be allowed after first dosing. All herbal or traditional Chinese medicines (e.g., St. John's Wort), within the 14 days prior to receiving the first dose of SM17, and continuing use if applicable, will be reviewed by the PI and the Medical Monitor. Written documentation of this review and acknowledgment is required for subject participation.
19. Has tattoo(s) or scarring at/or near the site of infusion or any other condition which may interfere with infusion site examination, in the opinion of the PI or designee.
20. Has been on a diet incompatible with the on study diet, in the opinion of the PI or designee, within the 30 days prior to the first dosing.
21. Donated blood (including blood products) or experienced loss of blood ≥ 500 mL within 2 months of the screening visit; blood donation or loss of blood ≥ 200 mL within 1 month prior to the screening visit; or plan to donate blood during the study period.
22. Plasma donation within 7 days prior to the first dosing.
23. Donated bone marrow within the last 3 months prior to the first dosing.
24. Will not be available for protocol-required study visits or procedures, to the best of the subject and PI or designee's knowledge.
25. Has any kind of disorder that, in the opinion of the PI or designee, may compromise the ability of the subject to give written informed consent and/or to comply with all required study procedures.
26. Is unwilling to avoid rigorous exercise for at least 48 hours prior to first dosing.
27. Is unwilling to avoid caffeinated beverages for at least 4 hours prior to first dosing.
28. Is receiving or has received any investigational drug (or is currently using an investigational device) within 30 days or 5 half-lives (whichever is longer) prior to the screening visit. The 30-day window (or 5 half-lives) will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to the screening visit of the current study.
29. Is receiving or has received any biologics within 90 days or until the expected PD effect has returned to baseline (whichever is longer) prior to the screening visit. The 90-day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to the screening visit of the current study.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-09-26 (Actual)

PRIMARY OUTCOMES:
Part A and Part B: Number of subjects with adverse events | Until Follow-up (FU) Visit/Early Termination (ET) Visit (14 and 28 days post-last dose)
  To evaluate the safety and tolerability of intravenous doses of SM17 in healthy adult subjects.

SECONDARY OUTCOMES:
Pharmacokinetic parameters of SM17 in healthy subjects | 0-20 weeks
  Pharmacokinetic parameters of SM17 in healthy subjects: peak concentration (Cmax)

OTHER OUTCOMES:
Pharmacokinetic parameters of SM17 in healthy subjects | 0-20 weeks
  Pharmacokinetic parameters of SM17 in healthy subjects: elimination half-life (T1/2)
Pharmacokinetic parameters of SM17 in healthy subjects: time to peak (Tmax) | 0-20 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion Lincoln, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xu G, Paglialunga S, Qian X, Ding R, Webster K, van Haarst A, Engel C, Hui CW, Lam LH, Li W, Wu WC, Rasmussen S, Hunt A, Leung SO. Evaluation of the safety, tolerability, pharmacokinetics and pharmacodynamics of SM17 in healthy volunteers: results from pre-clinical models and a first-in-human, randomized, double blinded clinical trial. Front Immunol. 2024 Dec 9;15:1495540. doi: 10.3389/fimmu.2024.1495540. eCollection 2024. PMID 39717777